CLINICAL TRIAL: NCT05605080
Title: Hemostatic and Analgesic Effect of Gel Foam and Gauze With Bosmin After Anal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, MD, PhD, Chief of Colorectal Surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202209015
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hemorrhoids; Anal Fistula
MeSH Terms: conditions — Hemorrhoids; Rectal Fistula | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Gelfoam as hemostatic agent after surgery (Experimental): Use Gelfoam as hemostatic agent after surgery.
  Interventions: Device: Gelfoam
- Gauze with Bosmin as hemostatic agent after anal surgery (Active Comparator): Use gauze with Bosmin as hemostatic agent after anal surgery
  Interventions: Other: Bosmin gauze

INTERVENTIONS:
Device: Gelfoam — Use Gelfoam as a hemostatic agent after anal surgery.
  Arms: Gelfoam as hemostatic agent after surgery
Other: Bosmin gauze — Use bosmin gauze as a hemostatic agent after anal surgery.
  Arms: Gauze with Bosmin as hemostatic agent after anal surgery

SUMMARY:
To evaluate the hemostatic and analgesic effect of using gauze with Bosmin or Gelfoam after anal surgery.

DETAILED DESCRIPTION:
Hemorrhoidectomy and fistulotomy these two types of anal surgery are common surgeries in colon and rectal surgery division in Shuang Ho hospital. For these patients underwent surgical treatment, some surgeons used gauze with Bosmin for hemostasis and analgesia after surgery, and other surgeons used Gelfoam. These choices were often determined by surgeon's personal preference according to their experiences. Shuang Ho hospital has top three quantity of hemorrhoidectomy in Taiwan. So, a randomized controlled trial is conducted to evaluate the difference between hemostatic agents use after anal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo conventional hemorrhoidectomy or stapled hemorrhonidpexy are include.
* Patients who undergo fistulectomy or fistulotomy are include.

Exclusion Criteria:

* Emergency operation
* Patients with colorectal cancer
* Liver cirrhosis
* Patients with coagulopathy
* Patients with HIV infection

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 0-7 days
  Record maximum pain score (visual analog scale, 0-10) from post-operative day 0 to day 7.
Analgesic agent use | 0-7days
  Daily consumption of oral analgesics from post-operative day 0 to day 7

SECONDARY OUTCOMES:
Incidence of post-operative bleeding | 0-30 days
  Postoperative delayed bleeding was defined as (1) when the bleeding required surgical intervention or (2) when hospital re-admission was warranted after patient discharge.
Incidence of urinary retention | 0-7 days
  Urinary retention was defined as patients requiring Foley catheterization during the hospital stay
Incidence of surgical site infection | 0-30 days
  Surgical site infection was defined as hospital admission for infection management or need for surgical intervention to manage the wound.

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Cheng Chang, MD, PHD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets used in this study can be obtained from the investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: data is available as the study is complete and for 12 month period
Access Criteria: will be shared upon request